CLINICAL TRIAL: NCT00810147
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, Pharmacodynamic and Pharmacokinetic Effects of BMS-708163 in the Treatment of Patients With Mild to Moderate Alzheimer's Disease
Brief Title: A Phase II, Multicenter, Double Blind, Placebo-Controlled Safety, Tolerability Study of BMS-708163 in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN156-013; EUDRACT: 2008-005929-11
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — BMS 708163

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- A1 (Active Comparator)
  Interventions: Drug: BMS-708163
- A2 (Active Comparator)
  Interventions: Drug: BMS-708163
- A3 (Active Comparator)
  Interventions: Drug: BMS-708163
- A4 (Active Comparator)
  Interventions: Drug: BMS-708163
- A5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-708163 — Capsules, Oral, 25 mg, once daily, 24 weeks
  Arms: A1
Drug: BMS-708163 — Capsules, Oral, 50 mg, once daily, 24 weeks
  Arms: A2
Drug: BMS-708163 — Capsules, Oral, 100 mg, once daily, 24 weeks
  Arms: A3
Drug: BMS-708163 — Capsules, Oral, 125 mg, once daily, 24 weeks
  Arms: A4
Drug: Placebo — Capsules, Oral, 0 mg, once daily, 24 weeks
  Arms: A5

SUMMARY:
The purpose of this study is to determine the safety and tolerability of BMS-708163 in patients with mild to moderate Alzheimer's disease over a treatment period of 12-weeks and the course of any potential effects during a 12-week wash-out period

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Mild to Moderate Alzheimer's disease (MMSE 16-26)
* 6 Month cognitive decline
* Stable marketed AD therapy x2 months or additional marketed AD therapy during study
* Score of <=4 on the Modified Hachinski Ischemia Scale
* CT results consistent with Alzheimer's disease
* Medically stable
* 6 years education
* Reliable study partner (caregiver)
* Must be able to swallow capsules

Exclusion Criteria:

* Premenopausal women
* Dementia due to other causes than Alzheimer's disease
* History of stroke
* Immunocompromised
* Active peptic ulcer, GI bleed, chronic inflammatory bowel disease, chronic diarrhea or past GI surgery that would impact drug absorption
* Unstable Vitamin B-12 deficiency
* Hematologic or solid malignancy within 5 years
* Geriatric Depression Scale >= 6
* Unstable medical condition
* Alcohol or drug abuse history with 12-months of study entry
* Significant drug allergy
* Alzheimer's disease modification experimental therapy with 12 months of study entry
* Prisoners, compulsory psychiatric patients, or residents of nursing home or skilled nursing facility at entry
* Any other experimental therapy with 30-days of study entry

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Weekly for the first 12-weeks of the 24-Week dosing period (Baseline-Week-12) and every 2 weeks during the second 12-weeks of the 24-Week dosing period (Weeks 14-24) and during the subsequent 12-week washout period (Weeks 28, 32, & 36)

SECONDARY OUTCOMES:
Pharmacodynamics effects of Cerebral Spinal Fluid | Baseline, Week 12 and Week 24
Pharmacodynamics effects of the Alzheimer's Disease Assessment Scale - Cognitive Subscale | Baseline, Week 12, Week 24 and Week 36
Pharmacodynamics effects of the Alzheimer's Disease Collaborative Study - Activities of Daily Living scale | Baseline, Week 12, Week 24 and Week 36
Pharmacodynamics effects of the Global clinical impression as assessed with the Clinical Dementia Rating-Sum of Boxes | Baseline, Week 12, Week 24 and Week 36
Characterize Pharmacodynamics/Pharmacokinetics effects of the plasma exposure of BMS-708163 and variability in a population with Alzheimer's disease | Baseline, Week 12 and Week 24
Characterize Pharmacodynamics/Pharmacokinetics effects in refining the Pharmacokinetics/Pharmacodynamics model with Phase 2 data | Baseline, Week 12 and Week 24
Characterize Pharmacodynamics/Pharmacokinetics effects by exploring correlations between exposure, biomarkers, and clinical effects | Baseline, Week 12 and Week 24
Characterize Pharmacodynamics/Pharmacokinetics effects by exploring Pharmacokinetics variability, including the correlation between polymorphisms of CYP enzymes | Baseline, Week 12 and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (41):
- United States (35):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - 21st Century Neurology, Phoenix, Arizona
  - Banner Alzheimer'S Institute, Phoenix, Arizona
  - Sun Health Research Institue, Sun City, Arizona
  - Margolin Brain Institute, Fresno, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Pacific Institute For Medical Research, Inc., Los Angeles, California
  - Mary S. Easton Center, Los Angeles, California
  - Pacific Research Network, Inc, San Diego, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Meridien Research, Brooksville, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Md Clinical, Hallandale, Florida
  - Compass Research, Llc, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Usf Suncoast Alzheimer'S And Gerontology Center, Tampa, Florida
  - Center For Clinical Trials, Venice, Florida
  - Indiana University Medical Center, Indianapolis, Indiana
  - Four Rivers Clinical Research, Inc, Paducah, Kentucky
  - Memory Enhancement Center Of Amercia, Inc., Eatontown, New Jersey
  - Global Medical Institutes, Llc, Princeton, New Jersey
  - Columbia University, New York, New York
  - University Of Rochester, Rochester, New York
  - Richard H. Weisler, Md, Pa & Associates, Raleigh, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Neurology & Neuroscience Center Of Ohio, Toledo, Ohio
  - Tulsa Clinical Research, Llc, Tulsa, Oklahoma
  - Professional Neurological Associates, Pc, Dunmore, Pennsylvania
  - The Clinical Trial Center Llc, Jenkintown, Pennsylvania
  - R.I. Mood & Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - The University Of Texas, Dallas, Texas
  - Dean Foundation For Health Research & Education, Middleton, Wisconsin
- Local Institution, Odense, Denmark
- Finland (2):
  - Local Institution, Kuopio
  - Local Institution, Turku
- Sweden (3):
  - Local Institution, Malmo
  - Local Institution, Mölndal
  - Local Institution, Stockholm

REFERENCES:
- [Derived] Coric V, van Dyck CH, Salloway S, Andreasen N, Brody M, Richter RW, Soininen H, Thein S, Shiovitz T, Pilcher G, Colby S, Rollin L, Dockens R, Pachai C, Portelius E, Andreasson U, Blennow K, Soares H, Albright C, Feldman HH, Berman RM. Safety and tolerability of the gamma-secretase inhibitor avagacestat in a phase 2 study of mild to moderate Alzheimer disease. Arch Neurol. 2012 Nov;69(11):1430-40. doi: 10.1001/archneurol.2012.2194. PMID 22892585
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx